CLINICAL TRIAL: NCT06565351
Title: Feasibility of Replacing 99mTc-DTPA GFR Measurements With eGFR From s-Cystatin C in Individuals With Spinal Cord Injuries
Brief Title: S-cystatin C vs.Injection Clearance Measurements to Estimate Kidney Function in Patients With Spinal Cord Injuries
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulrik Bjoern Andersen, Senior Consultant, Rigshospitalet, Denmark
Other Study IDs: Rigshospitalet; Glostrup
Record Dates: First submitted 2024-08-16; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries; Renal Failure
Keywords: spinal cord injury; renal Failure; GFR; Glomerular filtration rate; DTPA clearance; Cystatin C; eGFR
MeSH Terms: conditions — Spinal Cord Injuries; Renal Insufficiency | interventions — Cystatin C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Cord Injury Individuals: 248 individuals with spinal cord injury and neurogenic bladder dysfunction, coming to routine controls of the renal function. Glomerular filtration rate (GFR) was measured by 99mTc-DTPA clearance and estimated by eGFR from creatinine and Cystatine C
  Interventions: Other: eGFR estimated from creatinine and cystatin C

INTERVENTIONS:
Other: eGFR estimated from creatinine and cystatin C — eGFR estimated from creatinine and cystatin C was compared to GFR measured by 99mTc-DTPA clearance (gold standard)

SUMMARY:
* In individuals with spinal cord injury (SCI) kidney function defined as Glomerular Filtration Rate (GFR) is monitored by injection of e.g.99mDTPA and subsequent blood sampling (DTPA-clearance)
* GFR calculated from plasma samples of the endogenous substance s-Cystatin C (eGFR cystatin C) was compared to DTPA-clearance in 248 individuals with SCI.
* It is concluded that eGFR based on plasma s-cystatin C can replace the more tedious 99mDTPA-clearance procedures in individuals with SCI

ELIGIBILITY:
Inclusion Criteria:

Neurogenic bladder dysfunction due to spinal cord injury

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 248 consecutive individuals with neurogenic bladder dysfunction due to spinal cord injury coming to routine control of their kidney function every 2-3 years according to international guidelines
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Estimated clearance of Cystatin C (eGFR cystatin C) | through study period (2 years)
  The estimated clearance of cystatin (eGFR) C is calculated from s-cystatin C and the age and height and weight of the individual. It is corrected for Body Surface area. In this study it is compared to the Gold Standard examination DTPA-clearance

SECONDARY OUTCOMES:
Test/ retest variability of eGFR cystatin C | Up to three months
  Blood samples for determination of Cystatin C is taken twice within maximally three months, to determine the repeatability of eGFR cystatin C
Long term repeatability of eGFR cystatin C | Up to three years
  Blood samples for determination of cystatin C is taken twice with an interval of two-three years to determine long term repeatability. This is compared to simultaneously acquired measurements of DTPA-clearance

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik B. Andersen, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Dept. of Clinical Physiology and Nuclear Medicine, Copenhagen University Hospital, Rigshospitalet; Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers. Data or samples shared will be coded, with no personal health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 9-24 months after publication
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)